CLINICAL TRIAL: NCT01272492
Title: Infant Nutrition: Evaluation of an Educational Touchscreen Computer Program for Use in a Spanish-speaking Population of Caregivers of Young Children (APA Phase II)
Brief Title: Infant Nutrition: Evaluation of an Educational Touchscreen Computer Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Maryland (Other); Academic Pediatric Association (Industry)
Responsible Party: Darcy Thompson MD MPH, Johns Hopkins School of Medicine
Model: Parallel | Purpose: Prevention
Other Study IDs: NA_00035707
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2010-06

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Computer Use (Experimental): Participants use the computer with the infant/toddler nutrition/feeding education modules
  Interventions: Other: Computer Use
- Control (No Intervention): Only answers survey questions.

INTERVENTIONS:
Other: Computer Use — Participants use the computer with the 5 modules on infant/toddler feeding/nutrition
  Arms: Computer Use

SUMMARY:
The investigators are recruiting participants for a randomized controlled trial to evaluate the usability and educational value of a nutrition education touchscreen computer program targeting Spanish-speaking Latina caregivers of children 2 and under.

Participants will be randomized to the intervention group - use the computer program and the control group - do not use the program. They will be asked basic demographic questions, nutrition knowledge questions and computer users will be asked usability questions.

Objectives are

1. Evaluate the subjective and objective usability of the touchscreen computer.
2. Determine whether health knowledge on nutrition topics is enhanced through the use of the computer modules.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a child 2 and under in their care 2. Consider themselves Latina 3. Are Spanish-speaking

Exclusion Criteria:

Exclude if child has major medical issues interfering with feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's medical Practice, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Thompson DA, Joshi A, Hernandez RG, Bair-Merritt MH, Arora M, Luna R, Ellen JM. Nutrition education via a touchscreen: a randomized controlled trial in Latino immigrant parents of infants and toddlers. Acad Pediatr. 2012 Sep-Oct;12(5):412-9. doi: 10.1016/j.acap.2012.03.020. Epub 2012 Jun 7. PMID 22682718